CLINICAL TRIAL: NCT07376200
Title: An I-phase Clinical Trial Evaluating the Safety, Tolerability, Pharmacokinetic/Pharmacodynamic Characteristics of a Single Dose of HEC-151 Injection in Healthy Chinese Participants in a Single-center, Randomized, Placebo (Single-blind) and Positive Control (Open-label) Study
Brief Title: Single-ascending Dose Study of HEC-151 Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEC-151-DM-101
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Healthy Adult Male
Keywords: HEC-151 Injection
MeSH Terms: interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant
Masking Description: HEC-151 Injection, Insulin Degludec, placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEC-151 Injection and placebo (Experimental): The participants received an abdominal subcutaneous HEC-151 Injection or a placebo in the morning of Day 1.
  Interventions: Drug: HEC-151 Injection and placebo
- Insulin Degludec (Active Comparator): The participants received an abdominal subcutaneous injection of Insulin Degludec in the morning of Day 1.
  Interventions: Drug: Degludec insulin

INTERVENTIONS:
Drug: HEC-151 Injection and placebo — Subcutaneous injection in the abdominal area
  Arms: HEC-151 Injection and placebo
Drug: Degludec insulin — Subcutaneous injection in the abdominal area
  Arms: Insulin Degludec

SUMMARY:
Evaluate the safety, tolerability, PK/PD and immunogenicity characteristics of a single subcutaneous HEC-151 Injection solution in healthy participants

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the trial and sign the informed consent form, understanding and abiding by the research procedures;
2. When signing the informed consent form, men aged 18-45 years old (including the boundary value) are eligible;
3. During the screening process, male subjects with a body weight of ≥ 50 kg and a body mass index (BMI) of ≥ 19.0 and ≤ 24.0 kg/m2 are included;
4. Normal glucose tolerance [3.9 mmol/L < fasting blood glucose (FPG) < 6.1 mmol/L, and 2-hour post-glucose tolerance test (OGTT) blood glucose after sugar intake < 7.8 mmol/L];
5. Normal results of insulin release test (IRT), or abnormal results but judged by the researcher to have no clinical significance;
6. Glycated hemoglobin (HbA1c) < 5.7%;
7. During the study period, there are no plans for reproduction, sperm collection, or sperm donation, and are willing to take effective contraceptive measures throughout the study period until 3 months after the administration of the investigational drug.

Exclusion Criteria:

1. Participants with abnormal medical histories or surgical histories judged clinically significant by the researchers, or currently suffering from any diseases in the endocrine system, blood system, cardiovascular system, respiratory system, digestive system, urinary system, immune system, nervous system, etc. that are judged clinically significant by the researchers, or any other diseases or physiological conditions that can significantly affect the absorption, distribution, metabolism or excretion of the drugs;
2. Participants who have a known severe allergic history or are allergic to the test drugs and any of their components;
3. Participants who had severe trauma or undergone surgery within 90 days before the screening, or plan to undergo major surgery during the study;
4. Participants who have a history of hypoglycemia or hyperglycemia within 90 days before the screening, or have a family history of diabetes (first-degree direct relatives);
5. Participants who have donated blood or suffered significant blood loss (≥ 400 mL) within 90 days before the screening, or plan to donate blood during the study;
6. Participants who have acute diseases or concurrent medication use from the signing of the informed consent form to the first administration of the drug;
7. Participants whose vital signs, physical examination, laboratory tests, electrocardiogram, chest X-ray examination, etc. results are abnormal and judged by the researchers to have clinical significance;
8. Participants whose test results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV), combined human immunodeficiency virus antigen antibody (HIV), or syphilis spirochete antibody (TP) are positive;
9. Participants who have a history of drug abuse or drug use, or whose urine drug screening is positive before the screening;
10. Participants who have used any prescription drugs, Chinese herbal medicines, over-the-counter drugs, health supplements (except for regular supplementary vitamins and calcium) within 30 days before the screening;
11. Participants who have participated in any clinical research of drugs or devices (defined as receiving the test drugs or devices) within 90 days before the screening;
12. Participants who have received any vaccine within 30 days before the screening, or plan to receive any type of vaccine during the study;
13. Participants who smoke more than 5 cigarettes per day within 90 days before the screening, or cannot comply with the smoking prohibition rule during the study;
14. Participants who frequently drink alcohol, that is, consuming more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of 40% alcohol spirits or 150 mL of wine), or have a positive alcohol breath test; or who cannot comply with the alcohol prohibition rule during the study;
15. Participants who consume excessive tea, coffee and/or caffeine-rich beverages (more than 8 cups, 1 cup ≈ 250 mL) or food (such as chocolate) every day within 90 days before the screening, or during the study;
16. Participants who have used special diets (including dragon fruit, mango, pomelo, etc.) and/or xanthine diet (salmon, sardines, liver, kidney, etc.) or have other factors affecting drug absorption, distribution, metabolism, and excretion before the signing of the informed consent form to the use of the test drugs, or who cannot comply with the prohibition of eating during the study;
17. Participants who have had significant changes in diet or exercise habits within 90 days before the screening, or have engaged in intense exercise before the signing of the informed consent form to the use of the test drugs, or cannot stop during the study;
18. Participants who have difficulty in venous blood collection, or cannot tolerate venipuncture, or have a history of fainting or hematemesis;
19. Participants who, in the researcher's opinion, have other factors that are not suitable for participating in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Estimated)
Dates: Start 2026-03-11 (Estimated); Primary Completion 2026-09-05 (Estimated); Study Completion 2026-09-27 (Estimated)

PRIMARY OUTCOMES:
Adverse event | From Day1 to Day36
  Frequency, type and severity of adverse events/serious adverse events.
Electrocardiogram parameter（Heart rate） | From Day1 to Day36
  Evaluation the heart rate of electrocardiogram parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Electrocardiogram parameter（PR interval） | From Day1 to Day36
  Evaluation the PR interval of electrocardiogram parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Electrocardiogram parameter（QTcF interval） | From Day1 to Day36
  Evaluation the QTcF interval of electrocardiogram parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Electrocardiogram parameter(QRS interval) | From Day1 to Day36
  Evaluation the QRS interval of electrocardiogram parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Vital signs parameter（Body temperature） | From Day1 to Day36
  Evaluation the body temperature of vital signs parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Vital signs parameter（Blood pressure） | From Day1 to Day36
  Evaluation the blood pressure of vital signs parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Vital signs parameter（Pulse） | From Day1 to Day36
  Evaluation the pulse of vital signs parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.
Vital signs parameter（Respiration） | From Day1 to Day36
  Evaluation the respiration of vital signs parameters, and summarize the baseline data, post-administration data, and the changes from baseline after administration for each visit and treatment group.

SECONDARY OUTCOMES:
Cmax | From Day1 to Day36
  Evaluate the pharmacokinetic effects of HEC-151 Injection in healthy participants.
AUC0-t | From Day1 to Day36
  Evaluate the pharmacokinetic effects of HEC-151 Injection in healthy participants.
Tmax | From Day1 to Day36
  Evaluate the pharmacokinetic effects of HEC-151 Injection in healthy participants.
T1/2 | From Day1 to Day36
  Evaluate the pharmacokinetic effects of HEC-151 Injection in healthy participants.
CL/F | From Day1 to Day36
  Evaluate the pharmacokinetic effects of HEC-151 Injection in healthy participants.
GIRmax | From Day1 to Day36
  Evaluate the Pharmacodynamics effects of HEC-151 Injection in healthy participants.
tGIRmax | From Day1 to Day36
  Evaluate the Pharmacodynamics effects of HEC-151 Injection in healthy participants.
AUCGIR | From Day1 to Day36
  Evaluate the Pharmacodynamics effects of HEC-151 Injection in healthy participants.
ADA（Anti-Drug Antibody） | From Day1 to Day36
  Evaluate the Immunogenic characteristics of HEC-151 Injection in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 9, Shuangxing Avenue,, Bishan, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No